CLINICAL TRIAL: NCT02630472
Title: Efficacy and Safety of Adjuvant Topical Irrigation in the Treatment of Acute Exacerbation of Chronic Rhinosinusitis Following Functional Endoscopic Sinus Surgery (FESS)
Brief Title: Topical Irrigation Therapy for CRS
Acronym: QSIND
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional decision
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 821731
Record Dates: First submitted 2015-12-09; First posted 2015-12-15 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Rhinitis; Sinusitis
MeSH Terms: conditions — Rhinitis; Sinusitis | interventions — Quinine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinine Sulfate (Experimental): Each study participant randomized into the experimental arm will receive 28 tubes with 1mg/ml (6 mls total) of quinine sulfate, as well as 28 3cc syringes with the mucosal atomizing devices. The solutions will be supplied in light-protected tubes. Patients will apply 3 mls of quinine sulfate to each nostril twice per day. Thus the patients will be exposed to a maximum of 12mls or 12.0 mg of quinine per day.
  The Investigational Drug Service (IDS) will prepare and record the distribution of the irrigant. The Clinical Research Coordinator or Clinical Research Nurse will pick up the solutions and will demonstrate the application to the subject. The application of the solution is exactly the same as if the study subject were to irrigate with regular saline as part of their daily regimen for chronic rhinosinusitis.
  Interventions: Drug: Quinine Sulfate
- Placebo (Placebo Comparator): The placebo arm will be spiked with Sucrose Octaacetate which has a bitter taste, but does not stimulate sinonasal nitric oxide production.
  Each study participant will receive 28 tubes with 0.5mg/ml sucrose octaacetate, as well as 28 3cc syringes with the mucosal atomizing devices. The solutions will be supplied in light-protected tubes.
  The placebo arm will mirror the experimental arm exactly, except for the treatment solution contained in the vials.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quinine Sulfate — Our plan is to first study quinine against saline to determine efficacy and safety. The vast majority of patients with rhinosinusitis utilize low pressure / high volume (240mls) sinonasal lavage to cleanse the sinonasal cavity. The patients will be exposed to a maximum of 12mls or 12.0 mg of quinine. In standard tonic water, quinine is 8.3mg/100mls and thus an 8oz glass of Canada Dry tonic water has 19.6mg of quinine. Thus, the maximum systemic exposure in our study (assuming ingestion of the total nasal administration) is less than drinking one glass of tonic water / day. To put this in context, the therapeutic range of quinine to treat malaria is 10mg/kg true ileal digestibility (TID) (2100mg for a 70kg individual) nearly 200 X the dose the investigators are proposing.
  Arms: Quinine Sulfate
Drug: Placebo — In order to blind the participants to which arm they have been randomized into, the placebo arm will contain saline solution spiked with 0.5 mg/ml sucrose octaacetate. This solution will produce a bitter flavor similar to the one produced by quinine. There is no evidence that sucrose octaacetate produces nitric oxide production in the sinonasal cavity, nor is there evidence that it has any side effects (it is used to wean babies off of pacifiers) so the investigators feel it is an effective and safe option for a placebo.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the physiologic response of quinine-saline irrigations for acute exacerbation of uncomplicated chronic rhinosinusitis following endoscopic sinus surgery. Subjects who have previously had functional endoscopic sinus surgery with acute exacerbation of chronic rhinosinusitis will be randomized to either a quinine-saline or saline-placebo arm. The investigators will measure baseline and follow-up clinical and quality-of-life outcomes for both arms, and then compare the groups at the end of the study period. The investigators' hypothesis is that the participants in the quinine sulfate arm will perform better on all measures as compared to the control arm.

DETAILED DESCRIPTION:
Overall Objectives:

To evaluate the physiological differences between quinine-saline irrigations vs. saline-placebo irrigations for acute exacerbation of uncomplicated chronic rhinosinusitis following endoscopic sinus surgery. A secondary objective is to determine if the use of quinine is efficacious as an alternative therapy to treat bacterial rhinosinusitis.

Background:

Sinusitis is a common disorder accounting for an estimated 13 million physician office visits in the United States each year. The aggregated cost of sinusitis is approximately $8 billion annually, affecting an estimated 16% of the population in the United States. Despite multiple attempted treatments, including an estimated 550,000 surgeries per year, the disease continues to be a major health problem, both in expenditures and poor quality of life. Recent analysis of data from the National Ambulatory Medical Care Survey and the National Hospital Ambulatory Medical Care Survey from 2006 to 2010 showed that rhinosinusitis accounted for more outpatient antibiotic prescriptions in adults than any other diagnosis.

Chronic rhinosinusitis (CRS) represents a considerable subset of this population and accounts for a significant portion of expenditures and the vast majority of surgeries. It is defined as signs and symptoms of sinusitis lasting more than 12 weeks. Unlike the organisms responsible for acute rhinosinusitis, difficult to treat bacteria such as Pseudomonas aeruginosa, Staphylococcus aureus and Stenotrophomonas multiformia are often offending pathogens in CRS. Their prevalence increases in those patients who have already had sinus surgery and continue to get recurring sinus infections. Staph aureus and gram-negative organisms have been shown to account for roughly 60% of infections in those patients who have previously undergone endoscopic sinus surgery. Due to increasing drug resistance as well as the potential for biofilm formation, there has been an increasing pressure from both patients and clinicians alike to develop alternative treatments to systemic antibiotics. One commonly used alternative in patients who have had previous sinus surgery is topical saline irrigation with and without other topical preparations. Topical irrigations have much greater paranasal sinus penetration in post surgical patients. Commonly used topical preparations include: saline alone or saline mixed with mupirocin, gentamicin, tobramycin, ceftazadine, betadine, manuka honey, baby shampoo, budesonide or mometasone.

The investigators have recently identified a novel arm of upper airway innate immunity mediated by bitter taste receptors. When a subset of airway bitter taste receptors are activated they stimulate the respiratory epithelium to generate nitric oxide, an important component of sinus innate immunity that increases mucociliary clearance as well as diffuses into the mucus where it is bactericidal. A topical therapy to activate these taste receptors may help the sinuses clear infections through this natural innate defense mechanism. While the investigators have identified multiple bitter compounds that stimulate this response, quinine piqued our interest as it activates multiple bitter taste receptors and has already been used in the human nose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone Functional Endoscopic Sinus Surgery (FESS)
2. Purulent drainage on nasal endoscopy
3. Male or female subjects, 18 years of age or older
4. Patients seen at the Dept. of Otorhinolaryngology clinic at Hospital of the University of Pennsylvania (HUP), a tertiary care clinic

Exclusion Criteria:

1. Pregnant women
2. Immunocompromised patients
3. Granulomatous diseases with rhinologic manifestations (Wegner's, Sarcoid, Churg-Strauss)
4. Primary ciliary dyskinesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Quinine Sulfate: Each study participant randomized into the experimental arm will receive 28 tubes with 1mg/ml (6 mls) of quinine sulfate, as well as 28 3cc syringes with the mucosal atomizing devices. The solutions will be supplied in light-protected tubes. Patients will apply 3 mls of quinine sulfate to each nostril twice per day. Thus the patients will be exposed to a maximum of 12mls or 12.0 mg of quinine per day.
  The Investigational Drug Service (IDS) will prepare and record the distribution of the irrigant. The Clinical Research Coordinator or Clinical Research Nurse will pick up the solutions and will demonstrate the application to the subject. The application of the solution is exactly the same as if the study subject were to irrigate with regular saline as part of their daily regimen for chronic rhinosinusitis.
  Quinine Sulfate: Our plan is to first study quinine against saline to determine efficacy and safety. The vast majority of patients with rhinosinusitis utilize low pressure
- Placebo: The placebo arm will be spiked with Sucrose Octaacetate which has a bitter taste, but does not stimulate sinonasal nitric oxide production.
  Each study participant will receive 28 tubes with 0.5mg/ml sucrose octaacetate, as well as 28 3cc syringes with the atomizing devices. The solutions will be supplied in light-protected tubes.
  The placebo arm will mirror the experimental arm exactly, except for the treatment solution contained in the vials.
  Placebo: In order to blind the participants to which arm they have been randomized into, the placebo arm will contain saline solution spiked with 0.5 mg/ml sucrose octaacetate. This solution will produce a bitter flavor similar to the one produced by quinine. There is no evidence that sucrose octaacetate produces nitric oxide production in the sinonasal cavity, nor is there evidence that it has any side effects (it is used to wean babies off of pacifiers) so the investigators feel it is an effective and safe option for a plac
Period: Overall Study
Arm/Group | Quinine Sulfate | Placebo
Started | 10 | 0
Completed (Trial was discontinued due to physician priorities; no subjects completed the trial.) | 0 | 0
Not Completed | 10 | 0
Not completed — Physician Decision | 10 | 0

BASELINE CHARACTERISTICS:
Population: No data collected, no analysis performed.
Groups:
- Quinine Sulfate: Each participant in the experimental arm will receive 28 tubes with 1mg/ml (6 mls total) of quinine sulfate, as well as 28 3cc syringes with the atomizers. The solutions will be light-protected. Patients will apply 3 mls to each nostril twice per day. Patients will be exposed to 12.0 mg quinine per day.
  The Investigational Drug Service (IDS) will prepare and record the distribution of the irrigant. The Clinical Research Coordinator or Clinical Research Nurse will pick up the solutions and will demonstrate the application. The application of the solution is exactly the same as their daily regimen.
  Quinine Sulfate: Our plan is to first determine efficacy and safety. The patients will be exposed to a maximum of 12mls or 12.0 mg of quinine. Thus, the maximum systemic exposure in our study (assuming ingestion of the total nasal administration) is less than drinking one glass of tonic water / day. The therapeutic range of quinine to treat malaria is nearly 200 X the dose proposed.
- Placebo: The placebo arm will be spiked with Sucrose Octaacetate which has a bitter taste, but does not stimulate sinonasal nitric oxide production.
  Each study participant will receive 28 tubes with 0.5mg/ml sucrose octaacetate, as well as 28 3cc syringes with the mucosal atomizing devices. The solutions will be in light-protected tubes.
  The placebo arm will mirror the experimental arm exactly, except for the treatment solution contained in the vials.
  Placebo: In order to blind the participants to which arm they have been randomized into, the placebo arm will contain saline solution spiked with 0.5 mg/ml sucrose octaacetate. This solution will produce a bitter flavor similar to the one produced by quinine. There is no evidence that sucrose octaacetate produces nitric oxide production in the sinonasal cavity, nor is there evidence that it has any side effects (it is used to wean babies off of pacifiers) so the investigators feel it is an effective and safe option for a placebo.
- Total: Total of all reporting groups
Arm/Group | Quinine Sulfate | Placebo | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  | 6
  Male | 4 |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 10 |  | 10
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Microbiome Profile
Description: Pre and post treatment endoscopically-obtained sinonasal microbiologic cultures.
Time Frame: Baseline, Week 2, and Week 10
Population: This study was terminated. Partial data was collected and is misleading due to mis-dosing. This outcome measure was not evaluated.
Groups:
- Quinine Sulfate: Each study participant randomized into the experimental arm will receive 28 tubes with 1mg/ml (6 mls total) of quinine sulfate, as well as 28 3cc syringes with the mucosal atomizing devices. The solutions will be supplied in light-protected tubes. Patients will apply 3 mls of quinine sulfate to each nostril twice per day. Thus the patients will be exposed to a maximum of 12mls or 12.0 mg of quinine per day.
- Placebo: The placebo arm will be spiked with Sucrose Octaacetate which has a bitter taste, but does not stimulate sinonasal nitric oxide production.
  Each study participant will receive 28 tubes with 0.5mg/ml sucrose octaacetate, as well as 28 3cc syringes with the mucosal atomizing devices. The solutions will be supplied in light-protected tubes.
  Placebo: In order to blind the participants to which arm they have been randomized into, the placebo arm will contain saline solution spiked with 0.5 mg/ml sucrose octaacetate. This solution will produce a bitter flavor similar to the one produced by quinine. There is no evidence that sucrose octaacetate produces nitric oxide production in the sinonasal cavity, nor is there evidence that it has any side effects (it is used to wean babies off of pacifiers) so the investigators feel it is an effective and safe option for a placebo.
Arm/Group | Quinine Sulfate | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Lund-Kennedy Endoscope Score
Description: Pre and post treatment nasal endoscopy scored with a validated staging system for edema, -scored by an independent blind observer.
Time Frame: Baseline, Week 2, and Week 10
Population: This study was terminated. Partial data was collected and is misleading due to mis-dosing. This outcome was not measured.
Arm/Group | Quinine Sulfate | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in the 22-item Sinonasal Outcomes Test Score
Description: Pre and post treatment quality of life questionnaires (22-item Sinonasal Outcomes Test [SNOT-22]).
Time Frame: Baseline, Week 2, and Week 10
Population: as for outcome 2
Arm/Group | Quinine Sulfate | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Sniffin' Stick-12 Score
Description: Change in olfactory sense from baseline to week 10 will be measured using the Sniffin' Stick-12 system. Patients will smell each "sniffing pen" and record the smell they detect. A score between 0-12 will indicate olfactory sense.
Time Frame: Baseline, Week 2 and Week 10
Population: as for outcome 2
Arm/Group | Quinine Sulfate | Placebo
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Rescue Antibiotics
Description: The necessity for rescue oral antibiotics for persistent infection.
Time Frame: Week 2 and Week 10
Population: as for outcome 2
Arm/Group | Quinine Sulfate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year (approximately)
Description: This was a very low risk trial.
Arm/Group | Quinine Sulfate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 7/10 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinine Sulfate (N=10) | Placebo (N=0)
Worsening of sinus symptoms (Respiratory, thoracic and mediastinal disorders) | 7 (7) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT02630472/Prot_SAP_000.pdf